CLINICAL TRIAL: NCT05653284
Title: A Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of AK130 (TIGIT/TGF-β Bifunctional Fusion Protein) in Patients With Advanced Malignant Tumors
Brief Title: A Study of AK130 in Patients With Advanced Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK130-101
Record Dates: First submitted 2022-11-25; First posted 2022-12-16 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK130 (Experimental): Each subject will receive a single dose of AK130 every 3-week cycle (Q3W) or every 2-week cycle (Q2W). Participants may continue on study drug until unacceptable toxicity, or other withdrawal criteria is met.
  Interventions: Drug: AK130

INTERVENTIONS:
Drug: AK130 — IV infusion, specified dose on specified days.

SUMMARY:
A Phase I open label, dose-escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics and anti-tumor activity of AK130 (TIGIT/TGF-β bifunctional fusion protein) in patients with advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent and any locally required authorization obtained from the subject/legal representative.
2. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
3. Life expectancy ≥3 months.
4. Histologically or cytologically documented unresectable advanced or metastatic malignant tumor that has failed or intolerant of standard therapy, or for which no effective standard therapy is available.
5. Subject must have at least one measurable lesion according to RECIST Version1.1.
6. Adequate organ function.

Exclusion Criteria:

1. Any malignancy other than the disease under study within the past 3 years except for radically cured local cancers, such as basal cell skin cancer, carcinoma in situ of the cervix, or carcinoma in situ of breast.
2. Receipt of any anti-TIGIT, anti-TGF-β treatment.
3. Experienced a toxicity that led to permanent discontinuation of prior immunotherapy. All AEs while receiving prior immunotherapy have not completely resolved or resolved to Grade 1 prior to screening, required the use of additional immunosuppression other than corticosteroids.
4. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1，or to levels dictated in the inclusion/exclusion criteria, except toxicities not considered a safety risk (e.g., alopecia, neuropathy, or asymptomatic laboratory abnormalities).
5. Major surgical procedure within 4 weeks prior to the first dose of AK130 or still recovering from prior surgery.
6. History of organ transplant.
7. Known allergy or reaction to any component of the AK130 formulation. History of severe hypersensitivity reactions to other mAbs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of participants with adverse events (AEs) | From time ICF is signed until 90 days after last dose of AK130
Number of participants with DLTs | During the first four weeks of treatment with AK130

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 years
Disease control rate (DCR) | Up to approximately 2 years
Progression-free survival (PFS) | Up to approximately 2 years
Overall survival (OS) | Up to approximately 2 years
Duration of Response (DOR) | Up to approximately 2 years
Time to response (TTR) | Up to approximately 2 years
Maximum observed concentration (Cmax) of AK130 | From first dose of study drug through end of treatment (up to approximately 2 years)
  The endpoints for assessment of PK include serum concentrations of AK130 at different timepoints after AK130 administration.
Minimum observed concentration(Cmin) of AK130 | From first dose of study drug through end of treatment (up to approximately 2 years)
  The endpoints for assessment of PK include serum concentrations of AK130 at different timepoints after AK130 administration.
Area under the curve (AUC) of AK130 for assessment of pharmacokinetics | From first dose of study drug through end of treatment (up to approximately 2 years)
  The endpoints for assessment of PK include serum concentrations of AK130 at different timepoints after AK130 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of study drug through 30 days after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, Principal Investigator — The Cancer Hospital Affiliated to Shandong First Medical University
Locations (1):
- The Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China